CLINICAL TRIAL: NCT05890027
Title: Phenylephrine Versus Upper Eyelid Taping For Muller's Muscle Conjunctival Resection Evaluation
Brief Title: Phenylephrine Versus Eyelid Taping for Muller's Muscle-Conjunctival Resection (MMCR) Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Sara T. Wester, Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20230019
Record Dates: First submitted 2023-05-25; First posted 2023-06-05 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Ptosis, Eyelid
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phenylephrine and Eye Taping Group (Experimental): Participants in this group will initially have superior visual field testing done with the upper eyelid manually taped. Then, participants will have superior visual field testing done after receiving Phenylephrine 2.5% ophthalmic solution. Participants will be in each group for up to 60 minutes.
  Interventions: Drug: Phenylephrine Ophthalmic; Other: Eyelid Tape

INTERVENTIONS:
Drug: Phenylephrine Ophthalmic — One drop of Phenylephrine 2.5% ophthalmic solution to be administered to the eye with ptosis to evaluate for surgical repair.
Other: Eyelid Tape — Participants will have the affected eye with ptosis manually lifted using tape.

SUMMARY:
This research study aims to compare whether Phenylephrine 2.5% ophthalmic eye drop solution can serve as a better indicator of the effect of a drooping upper eyelid (ptosis) by covering part of the upper portion of the field of vision as compared to traditional use of tape to lift up the upper eyelid in the evaluation of patients for surgical upper eyelid repair.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with ptosis undergoing conjunctival Muller's muscle resection evaluation.
* Individuals who can tolerate and have no hypersensitivity to phenylephrine 2.5% ophthalmic solution.
* Individuals who can tolerate eye-drop medications.
* Individuals who are physically able to take a tangent screen visual field test.
* Age: Adults who can comprehend the instructions and procedures (18+ years old)

Exclusion Criteria:

- This study will not incorporate any of the following at-risk populations: adults unable to consent, individuals who are not yet adults, pregnant women, prisoners.

* This study will not include participants who refuse to consent.
* This study will not include participants who are too tired or unable to take a tangent screen visual field test (see Risk to Subjects).
* This study will not include individuals who may not be able to tolerate phenylephrine 2.5% ophthalmic solution.
* Specifically, those with a past medical history of bradycardia, hypotension, autonomic dysfunction, or severe cardiovascular disease
* This study will not include individuals who consume drugs contraindicated in phenylephrine use: Ergot Derivatives (Vasoconstrictive CYP3A4 Substrates), Iobenguane Radiopharmaceutical Products, Kratom, Lisuride, Monoamine Oxidase Inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara T Wester, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study used an eye-based unit of analysis, where each eye with ptosis served as an individual study unit. Participants with bilateral ptosis contributed two eyes to the study, while those with unilateral ptosis contributed one eye. This was a single-arm study in which all recruited eyes progressed sequentially through identical interventions and assessments as described in the Arm/Group Description.
Units Other Than Participants: eyes
Groups:
- All Study Participants: This study used an eye-based unit of analysis, where each eye with ptosis served as an individual study unit. Participants with bilateral ptosis contributed two eyes to the study, while those with unilateral ptosis contributed one eye. All affected eyes underwent identical interventions and assessments in a single arm, sequential design as outlined below.
  Study Protocol:
  Each eye with ptosis underwent the following sequential interventions and assessments:
  1. Baseline measurements: Superior visual field (SVF) testing and margin reflex distance 1 (MRD1) measurements were performed with the eyelid in its natural position.
  2. Eyelid taping intervention: The upper eyelid was manually elevated using adhesive tape, and SVF testing was repeated.
  3. Phenylephrine intervention: One drop of 2.5% phenylephrine ophthalmic solution was instilled into the affected eye, followed by both SVF testing and MRD1 measurements.
  The total duration for each participant was less than 60 minutes across all testing conditions.
  Post-Study Assessment:
  Following completion of all interventions, participants completed a satisfaction questionnaire using a 5-point Likert scale to evaluate their experience with both eyelid taping and phenylephrine administration.
Period: Overall Study
Arm/Group | All Study Participants
Started | 18; 32 eyes
Completed | 18; 32 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- All Study Participants: This study used an eye-based unit of analysis, where each eye with ptosis served as an individual study unit. Participants with bilateral ptosis contributed two eyes to the study, while those with unilateral ptosis contributed one eye. All affected eyes underwent identical interventions and assessments.
  Study Protocol:
  Each eye with ptosis underwent the following sequential assessments:
  1. Baseline measurements: Superior visual field (SVF) testing and margin reflex distance 1 (MRD1) measurements were performed with the eyelid in its natural position.
  2. Eyelid taping intervention: The upper eyelid was manually elevated using tape, and SVF testing was repeated.
  3. Phenylephrine intervention: One drop of 2.5% phenylephrine ophthalmic solution was instilled into the affected eye, followed by both SVF testing and MRD1 measurements.
  The total duration for each participant was less than 60 minutes across all testing conditions.
  Post-Study Assessment: Following completion of all interventions, participants completed a satisfaction questionnaire using a 5-point Likert scale to evaluate their experience with both eyelid taping and phenylephrine administration.
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
Age, Customized [Count of Participants; unit: Participants]
  >18 years old | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18
Baseline MRD1 [Mean (Standard Deviation); unit: mm] | 0.69 (0.95)
Baseline Superior Visual Field [Mean (Standard Deviation); unit: degrees] | 7.20 (2.72)

OUTCOME MEASURES:

1. Primary Outcome: Mean MRD1 After Phenylephrine
Description: Margin to Reflex Distance 1 measured at least ten minutes after administration of a single drop of 2.5% phenylephrine ophthalmic solution into the superior conjunctival fornix of the eye. Measured in mm.
Time Frame: 10 minutes after phenylephrine instillation.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
mm | 2.08 (0.91)

2. Primary Outcome: Mean Change in MRD1 Between Baseline and Phenylephrine
Description: Change in Margin to Reflex Distance 1 between the eye at baseline and after instillation of 2.5% phenylephrine ophthalmic solution. Measured in mm.
Time Frame: Baseline, 10 minutes after phenylephrine instillation.
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
mm | 1.38 [1.18 to 1.59]

3. Primary Outcome: Mean Superior Visual Field After Taping
Description: Degree of ptosis as measured by a tangent screen superior visual field test after taping of the upper eyelid.
Time Frame: Baseline, Within 1 minute after upper eyelid taping.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
degrees | 21.40 (2.69)

4. Primary Outcome: Mean Change in Superior Visual Field After Taping
Description: Mean Change in Superior Visual Field between the eye at baseline and after taping of the upper eyelid. Measured in degrees.
Time Frame: Baseline, Within 1 minute after upper eyelid taping.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
degrees | 14.20 (3.53)

5. Primary Outcome: Count of Eyes That Met Insurance Criteria After Taping
Description: Insurance SVF criteria for determining if ptosis is functionally significant are based on the absolute SVF height in primary gaze (a superior visual field of 30 degrees or less from fixation at baseline) and the difference in SVF demonstrated by taping of the upper eyelids (improvement of at least 12 degrees in the superior visual field compared to baseline).
  Here we assessed the count of units, with units being eyes, that demonstrated an improvement of at least 12 degrees in superior visual field between baseline and taping of the upper eyelid.
Time Frame: Baseline, Within 1 minute after upper eyelid taping.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
eyes
  Achieved min 12 degree improvement | 27
  Did not achieve min 12 degree improvement | 5

6. Primary Outcome: Mean Superior Visual Field After Phenylephrine
Description: Degree of ptosis as measured by a tangent screen superior visual field test ten minutes after the administration of a single drop of 2.5% phenylephrine ophthalmic solution into the superior conjunctival fornix of the eye.
Time Frame: 10 minutes after phenylephrine instillation.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
degrees | 22.27 (3.56)

7. Primary Outcome: Mean Change in Superior Visual Field After Phenylephrine
Description: Change in superior visual field between baseline and 10 minutes after instillation of phenylephrine ophthalmic solution. Measured in degrees.
Time Frame: Baseline, 10 minutes after phenylephrine instillation.
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
degrees | 15.07 (3.58)

8. Primary Outcome: Count of Eyes That Met Insurance Criteria After Phenylephrine
Description: Insurance SVF criteria for determining if ptosis is functionally significant are based on the absolute SVF height in primary gaze (a superior visual field of 30 degrees or less from fixation at baseline) and the difference in SVF demonstrated by taping of the upper eyelids (improvement of at least 12 degrees in the superior visual field compared to baseline).
  Here we assessed the count of units, with units being eyes, that demonstrated an improvement of at least 12 degrees in superior visual field between baseline and phenylephrine ophthalmic solution instillation.
Time Frame: Baseline, 10 minutes after phenylephrine instillation.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Number analyzed (eyes) | 32
eyes
  Achieved min 12 degree improvement | 28
  Did not achieve min 12 degree improvement | 4

9. Secondary Outcome: Mean Participant Satisfaction Score After Taping
Description: After completing the testing, participants completed a post-study questionnaire using a 5-point Likert scale (5=excellent, 4=good, 3=average, 2=poor, 1=very poor) to rate their satisfaction and overall experience with both upper eyelid taping and 2.5% phenylephrine ophthalmic solution instillation.
Time Frame: Baseline, Within 5 minutes after completing SVF testing after phenylephrine instillation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
score on a scale | 3.69 (0.59)

10. Secondary Outcome: Mean Participant Satisfaction Score After Phenylephrine
Description: as for outcome 9
Time Frame: Baseline, Within 5 minutes after completing SVF testing after phenylephrine instillation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
score on a scale | 4.38 (0.79)

11. Secondary Outcome: Mean Change in Participant Satisfaction Score Between Taping and Phenylephrine
Description: as for outcome 9
Time Frame: Baseline, Within 5 minutes after completing SVF testing after phenylephrine instillation.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
score on a scale | 0.69 [0.41 to 0.97]

ADVERSE EVENTS:
Time Frame: 1 year
Description: This eye-based study treated each ptotic eye as an individual unit. Bilateral ptosis participants contributed two eyes; unilateral ptosis participants contributed one eye. All eyes underwent identical sequential interventions and assessments in this single-arm study. Since all participants received the same intervention sequence, adverse events are reported under one arm: "all study participants."
Groups:
- All Study Participants: This study used an eye-based unit of analysis, where each eye with ptosis served as an individual study unit. Participants with bilateral ptosis contributed two eyes to the study, while those with unilateral ptosis contributed one eye. All affected eyes underwent identical interventions and assessments.
  Study Protocol:
  Each eye with ptosis underwent the following sequential assessments:
  1. Baseline measurements: Superior visual field (SVF) testing and margin reflex distance 1 (MRD1) measurements were performed with the eyelid in its natural position.
  2. Eyelid taping intervention: The upper eyelid was manually elevated using tape, and SVF testing was repeated.
  3. Phenylephrine intervention: One drop of 2.5% phenylephrine ophthalmic solution was instilled into the affected eye, followed by both SVF testing and MRD1 measurements.
  All recruited eyes progressed through all testing conditions (baseline, taping, and phenylephrine ophthalmic solution).
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/27/NCT05890027/Prot_SAP_000.pdf